CLINICAL TRIAL: NCT02417883
Title: Furosemide Stress Test as a Predictor of Tubular Atrophy and Interstitial Fibrosis in Patients With Chronic Kidney Disease
Brief Title: Furosemide Stress Test as a Predictor of Tubular Function in Chronic Kidney Disease
Acronym: FST-IFTA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, Chief of Nephrology Department, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PT15-920
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease
Keywords: Furosemide; Interstitial Fibrosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pulmonary Fibrosis | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Furosemide Stress Test (Experimental): Furosemide stress test will be perform to patients scheduled for kidney bipsy. The test consist in 1.5 miligrams per kilogram of weight of intravenous furosemide administration, along with urinary output follow up and measurement for 6 hours. The urinary output will be replaced intravenously with normal saline to avoid dehydration and/or hypotension.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Evaluate urinary excretion rate fo furosemide

SUMMARY:
In kidney diseases, tubule-interstitium has become much more relevant, as formerly only the glomerulus was considered to have the main importance. Kidney's tubular atrophy and interstitital fibrosis is now recognized as long term prognostic value. We aim to evaluate the function of the kidney's tubule-interstitium through furosemide excretion after intravenous administration of this drug, and correlate the rate of excretion of furosemide with interstitial fibrosis findings in scheduled kidney biopsy for patients with chronic kidney disease.

DETAILED DESCRIPTION:
All patients scheduled for kidney biopsy will be invited to participate in a standard isovolemic furosemide stress test before the biopsy procedure. The latter will consist in 1.5 miligrams per kilogram of weight of intravenous furosemide administration, with urinary output follow up and measurement. The urinary output will be replaced intravenously with normal saline to avoid dehydration and/or hypotension. A standard 5ml sample of blood will be taken before the test and aliquots of urine before and after furosemide administration will be frozen.

After completion of the formely mentioned test, patients will proceed to their scheduled kidney biopsy along with interventions considered appropiate by their attending physician.

Kidney biopsy sample will be examined by histopathology service and the degree of interstitial fibrosis will be described. The degree of fibrosis will be correlated with the degree furosemide excretion and urinary output.

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate (informed consent)
* Legal age or older
* An estimated glomerular filtration rate greater than 15ml/min/1.73m2, calculated by CKD-EPI.

Exclusion Criteria:

* Known Alergic reaction to furosemide
* Contraindication to kidney biopsy
* Patient already in renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Urinary Output | 6 hours
  Cuantify urinary output after furosemide administration

SECONDARY OUTCOMES:
Furosemide excretion rate | 6hrs
  Cuantify furosemide excretion in urine
Interstitial Fibrosis | 3 days
  Measure interstitial fibrosis in kidney biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, MD, Principal Investigator — Chief of the Nephrology Department
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Boor P, Ostendorf T, Floege J. Renal fibrosis: novel insights into mechanisms and therapeutic targets. Nat Rev Nephrol. 2010 Nov;6(11):643-56. doi: 10.1038/nrneph.2010.120. Epub 2010 Sep 14. PMID 20838416
- [Background] Burns WC, Kantharidis P, Thomas MC. The role of tubular epithelial-mesenchymal transition in progressive kidney disease. Cells Tissues Organs. 2007;185(1-3):222-31. doi: 10.1159/000101323. PMID 17587828
- [Background] Farris AB, Chan S, Climenhaga J, Adam B, Bellamy CO, Seron D, Colvin RB, Reeve J, Mengel M. Banff fibrosis study: multicenter visual assessment and computerized analysis of interstitial fibrosis in kidney biopsies. Am J Transplant. 2014 Apr;14(4):897-907. doi: 10.1111/ajt.12641. Epub 2014 Feb 20. PMID 24712330
- [Background] Farris AB, Colvin RB. Renal interstitial fibrosis: mechanisms and evaluation. Curr Opin Nephrol Hypertens. 2012 May;21(3):289-300. doi: 10.1097/MNH.0b013e3283521cfa. PMID 22449945
- [Background] van der Voort PH, Boerma EC, Pickkers P. The furosemide stress test to predict renal function after continuous renal replacement therapy. Crit Care. 2014 May 14;18(3):429. doi: 10.1186/cc13871. No abstract available. PMID 25033085
- [Result] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972
- [Derived] Rivero J, Rodriguez F, Soto V, Macedo E, Chawla LS, Mehta RL, Vaingankar S, Garimella PS, Garza C, Madero M. Furosemide stress test and interstitial fibrosis in kidney biopsies in chronic kidney disease. BMC Nephrol. 2020 Mar 6;21(1):87. doi: 10.1186/s12882-020-01721-z. PMID 32143585